CLINICAL TRIAL: NCT06490406
Title: Communication Practices to Develop the Health Literacy Competencies in Nursing Students: A Randomized Controlled Trial
Brief Title: Communication Practices to Develop the Health Literacy Competencies in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: sol-201900138441-tra
Record Dates: First submitted 2024-06-13; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Health Literacy; Competence; Nursing Students
Keywords: Health Communication; Formative feedback; Health Literacy; Randomized Controlled Trial; Simulation

STUDY DESIGN:
Intervention Model Description: This study is a parallel group-randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the data analyst will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (EG1) (Experimental): In addition to the usual training in communication skills, a systematic and digitalized guide will be used that included the "health literacy practices" qualified by Coleman et al. [10] as a training complement and self-assessment of its performance. They will also receive feedback from independent observers (according to the systematic guide).
  Interventions: Behavioral: Multimodal intervention (communication and education simulations) for EG1
- Control Group / Experimental Group 2 (CG / EG2) (No Intervention): The CG will receive the usual training (consisting of two weekly meetings of two hours each with seven sessions whose main topics were social skills for clinical interviews: opening and closing of the clinical interviews, non-verbal communication, active listening, empathy, helping relationship, giving information about the nature of the disease and rationality of the therapeutic measures, health education, and negotiation). Furthermore, throughout the course, they will self-assess their performance using the opening video recording without systematic guidance and they will receive feedback about their communication practices during this first performance.
  Thus, CG will receive the full intervention after being evaluated (post-test 1 assessment), becoming the delayed Experimental Group 2 (EG2)

INTERVENTIONS:
Behavioral: Multimodal intervention (communication and education simulations) for EG1 — In summary, students in EG1 received the following multimodal intervention flow: 1) Health communication training, 2) Structured educational simulation using standardized patients (SPs), and 3) simulation feedback and self-assessment using a systematic guide that included the "health literacy practices".
  Arms: Experimental Group 1 (EG1)

SUMMARY:
Communication is a key health literacy educational competency in the professional training of health providers. However, students often have difficulty in applying theoretical communication models to the reality of clinical practice. Multimodal interventions based on simulation models emerge as an essential element to overcome this gap. During the simulation training, students must be aware of their communication errors and the needs that patients share in a clinical interaction.

The aim is to evaluate the effectiveness of multimodal training, which incorporates a systematic feedback guide about the student's clinical interview simulation performance, as a training complement to classical education to improve health literacy competencies and clear communication practices in health sciences students.

A randomized controlled trial will be conducted on 82 second-year nursing students recruited from the University of Cadiz. The experimental and control groups will receive the same communication multimodal training except for the inclusion of feedback on key aspects of communication for health literacy, which the experimental groups only used. Students will be assessed through clinical interview simulations by external observers. Bivariate and inferential statistical analyses will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Second-year nursing students at the University of Cadiz enrolled in the Interpersonal Communication Skills subject.

Exclusion Criteria:

* Absence in training.
* Does not consent to participate in the study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical relationship during the healthcare process | 5 months
  Clinical relationship developed between a healthcare professional and a patient was measured through CICAA scale (pre-test, post-test 1, and post-test 2).
  The CICAA scale is a measure instrument designed to assess the clinical relationship (CR) developed between a health professional and a patient. It can be used to evaluate global or partial aspects of CR, is based on an external evaluation through observation of the interaction and can be used for teaching purposes. For all 29 items (scored 0, 1, 2), the minimum score is 0, and the maximum score is 58. The higher the score, the better the communication skills in the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Bas-Sarmiento, Ph.D., Principal Investigator — University of Cadiz
Locations (1):
- Faculty of Nursing, University of Cadiz, Algeciras, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available when the results of the study will be published.
Access Criteria: Data will be published in supplementary material or they will available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Cusatis R, Holt JM, Williams J, Nukuna S, Asan O, Flynn KE, Neuner J, Moore J, Makoul G, Crotty BH. The impact of patient-generated contextual data on communication in clinical practice: A qualitative assessment of patient and clinician perspectives. Patient Educ Couns. 2020 Apr;103(4):734-740. doi: 10.1016/j.pec.2019.10.020. Epub 2019 Oct 30. PMID 31744702
- [Background] Abdolrahimi M, Ghiyasvandian S, Zakerimoghadam M, Ebadi A. Antecedents and Consequences of Therapeutic Communication in Iranian Nursing Students: A Qualitative Research. Nurs Res Pract. 2017;2017:4823723. doi: 10.1155/2017/4823723. Epub 2017 Dec 13. PMID 29387487
- [Background] Sorensen K, Van den Broucke S, Fullam J, Doyle G, Pelikan J, Slonska Z, Brand H; (HLS-EU) Consortium Health Literacy Project European. Health literacy and public health: a systematic review and integration of definitions and models. BMC Public Health. 2012 Jan 25;12:80. doi: 10.1186/1471-2458-12-80. PMID 22276600
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Coleman CA, Hudson S, Maine LL. Health literacy practices and educational competencies for health professionals: a consensus study. J Health Commun. 2013;18 Suppl 1(Suppl 1):82-102. doi: 10.1080/10810730.2013.829538. PMID 24093348
- [Background] Coleman C, Hudson S, Pederson B. Prioritized Health Literacy and Clear Communication Practices For Health Care Professionals. Health Lit Res Pract. 2017 Jul 10;1(3):e91-e99. doi: 10.3928/24748307-20170503-01. eCollection 2017 Jul. PMID 31294254
- [Background] Karuranga S, Sorensen K, Coleman C, Mahmud AJ. Health Literacy Competencies for European Health Care Personnel. Health Lit Res Pract. 2017 Dec 11;1(4):e247-e256. doi: 10.3928/24748307-20171005-01. eCollection 2017 Oct. PMID 31294270
- [Background] Helitzer DL, Lanoue M, Wilson B, de Hernandez BU, Warner T, Roter D. A randomized controlled trial of communication training with primary care providers to improve patient-centeredness and health risk communication. Patient Educ Couns. 2011 Jan;82(1):21-9. doi: 10.1016/j.pec.2010.01.021. Epub 2010 Mar 12. PMID 20219315
- [Background] Toronto CE. Health Literacy Competencies for Registered Nurses: An e-Delphi Study. J Contin Educ Nurs. 2016 Dec 1;47(12):558-565. doi: 10.3928/00220124-20161115-09. PMID 27893919
- [Background] Yin HS, Jay M, Maness L, Zabar S, Kalet A. Health Literacy: An Educationally Sensitive Patient Outcome. J Gen Intern Med. 2015 Sep;30(9):1363-8. doi: 10.1007/s11606-015-3329-z. PMID 26173523
- [Background] MacLean S, Kelly M, Geddes F, Della P. Use of simulated patients to develop communication skills in nursing education: An integrative review. Nurse Educ Today. 2017 Jan;48:90-98. doi: 10.1016/j.nedt.2016.09.018. Epub 2016 Sep 28. PMID 27741440
- [Background] Zhang H, Yoong SQ, Dong YH, Goh SH, Lim S, Chan YS, Wang W, Wu XV. Using a 3-Phase Peer Feedback to Enhance Nursing Students' Reflective Abilities, Clinical Competencies, Feedback Practices, and Sense of Empowerment. Nurse Educ. 2023 Jan-Feb 01;48(1):E11-E16. doi: 10.1097/NNE.0000000000001294. Epub 2022 Sep 21. PMID 36137289
- [Background] Toronto CE, Weatherford B. Health Literacy Education in Health Professions Schools: An Integrative Review. J Nurs Educ. 2015 Dec;54(12):669-76. doi: 10.3928/01484834-20151110-02. PMID 26652801